CLINICAL TRIAL: NCT02124421
Title: Phase II Randomized Study: Cytoreductive Surgery (CRS) With/Without Carboplatin Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Followed by Adjuvant Chemotherapy as Initial Treatment of Ovarian, Fallopian Tube, & Primary Peritoneal Cancer
Brief Title: HOT: HIPEC in Ovarian Cancer as Initial Treatment
Acronym: CRS/HIPEC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC-2014-17
Record Dates: First submitted 2014-04-13; First posted 2014-04-28 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Ovarian Carcinoma; Fallopian Tube Carcinoma
Keywords: Ovarian cancer; Cytoreductive surgery; Hyperthermic Intraperitoneal chemotherapy; Systemic chemotherapy; Primary peritoneal carcinoma; Fallopian Tube cancer; Intraperitoneal chemotherapy; IV/IP chemotherapy; IV chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Cytoreduction Surgical Procedures; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Surveys and Questionnaires; Hyperthermic Intraperitoneal Chemotherapy; Carboplatin; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRS with adjuvant IV/IP chemotherapy (Active Comparator): Patients undergo cytoreductive surgery (CRS) alone with IV/IP combination adjuvant chemotherapy. Day 1: IV paclitaxel (135 mg/m2), day 2: IP cisplatin (75 mg/m2), and day 8: IP paclitaxel (60 mg/m2) given every 21 days for a total of 6 cycles. Standard of care treatment. Administration of quality of life questionnaires throughout study duration of follow-up
  Interventions: Procedure: Cytoreductive Surgery (CRS); Drug: Adjuvant Chemotherapy; Other: Questionnaire; Drug: Paclitaxel; Drug: Cisplatin
- CRS/HIPEC with adjuvant IV chemotherapy (Experimental): Cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC) administered using carboplatin for 90 minutes. Adjuvant systemic IV combination chemotherapy with carboplatin and paclitaxel (Carboplatin AUC 6, Paclitaxel 175mg/m2) will be given every 21 days for a total of 6 cycles. Administration of quality of life questionnaires throughout study duration of follow-up
  Interventions: Procedure: Cytoreductive Surgery (CRS); Drug: Adjuvant Chemotherapy; Other: Questionnaire; Procedure: Hyperthermic intraperitoneal chemotherapy; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Procedure: Cytoreductive Surgery (CRS) — Cytoreductive surgery
  Other Names: CRS
Drug: Adjuvant Chemotherapy — Six weeks post-surgery (CRS or CRS/HIPEC) standard combination chemotherapy will be administered every 21 days for 6 cycles
  Other Names: Post-operative chemotherapy; Systemic chemotherapy
Other: Questionnaire — Questionnaires designed to assess quality of life in ovarian cancer patients will be administered to study participants
  Other Names: FACT-O Questionnaire
Procedure: Hyperthermic intraperitoneal chemotherapy — Hyperthermic intraperitoneal chemotherapy with carboplatin, AUC=6
  Other Names: HIPEC
  Arms: CRS/HIPEC with adjuvant IV chemotherapy
Drug: Carboplatin — AUC=6 mg/mL/min IV (in the vein), on day 1. Repeat every 21 days for 6 cycles.
  Other Names: Paraplatin
  Arms: CRS/HIPEC with adjuvant IV chemotherapy
Drug: Paclitaxel — 175 mg/m2 IV (in the vein), day 1. Repeat every 21 days for 6 cycles
  Other Names: Taxol
  Arms: CRS/HIPEC with adjuvant IV chemotherapy
Drug: Paclitaxel — Day 1: paclitaxel 135 mg/m2 IV (in the vein). Repeat every 21 days for 6 cycles Day 8: paclitaxel 60 mg/m2 IP (intraperitoneal). Repeat every 21 days for 6 cycles
  Other Names: Taxol
  Arms: CRS with adjuvant IV/IP chemotherapy
Drug: Cisplatin — Day 2: cisplatin 75 mg/m2 IP (intraperitoneal). Repeat every 21 days for 6 cycles
  Other Names: CDDP
  Arms: CRS with adjuvant IV/IP chemotherapy

SUMMARY:
Community hospital based phase II (prospective randomized) study to evaluate the toxicity of cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) in newly diagnosed, otherwise untreated, advanced stage (stage III/IV) epithelial ovarian, fallopian tube, and primary peritoneal cancer.

DETAILED DESCRIPTION:
Primary endpoints:

* To assess the feasibility of recruitment
* Compare complication rates between the two study arms: CRS with HIPEC and CRS alone.

Secondary endpoints:

* To determine risk factors for morbidity and mortality
* Assess completion rate of 6 cycles of systemic chemotherapy
* To determine progression free survival at 24 months
* To determine overall survival at 1, 3, and 5 years
* Evaluate health related quality of life

Patients who meet study criteria will be randomized into one of two treatment arms: 1) cytoreductive surgery (CRS) with carboplatin-based hyperthermic intraperitoneal chemotherapy (HIPEC) followed by IV combination chemotherapy with carboplatin and paclitaxel or 2) cytoreductive surgery (CRS) alone followed by adjuvant intraperitoneal (IP) and IV chemotherapy with combination cisplatin and paclitaxel for newly diagnosed advanced stage (stage III/IV) ovarian, fallopian tube or primary peritoneal cancer. Both study arms will receive 6 cycles of adjuvant chemotherapy.

Twenty-four patients will undergo CRS with HIPEC performed by surgical and gynecologic oncologic surgeons at Mercy Medical Center, followed by systemic IV chemotherapy with carboplatin (AUC=6) and paclitaxel (175mg/m2) for 6 cycles postoperatively.

Twenty-four patients will undergo CRS only performed by surgical and gynecologic oncologic surgeons at Mercy Medical Center, followed by IV/IP chemotherapy with Day 1: IV paclitaxel (135 mg/m2), Day 2: IP cisplatin (75 mg/m2), and Day 8: IP paclitaxel (60 mg/m2) for 6 cycles postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation of ovarian, fallopian tube or primary peritoneal cancer
* Stage III/IV disease
* No prior treatment or significant surgery for the management of ovarian, fallopian tube, or primary peritoneal carcinoma; History of laparoscopic procedures to obtain diagnostic biopsies will be permitted in the study
* Histological confirmation
* Eastern Cooperative Oncology Group performance status 0-2 or Karnofsky performance status ≥ 70%
* ≤1 cm residual disease at the completion of the cytoreductive surgery (GOG criteria for optimally cytoreduction)
* Bone marrow function:

  1. Absolute neutrophil count (ANC) ≥1,000/mm3
  2. Platelets ≥100,000/mm3
  3. Hemoglobin ≥ 8.5 g/dL
* Renal function:

  1) Creatinine ≤1.5 times the upper limit of normal or a calculated creatinine clearance ≥60ml/min
* Hepatic function:

  1. Bilirubin ≤1.5 times upper limit of normal
  2. Alanine aminotransferase (ALT) ≤3 times upper limit of normal
  3. Aspartate aminotransferase (AST) ≤3 times upper limit of normal
* Blood coagulation parameters:

  1. Prothrombin time (PT) with International Normalized Ratio of ≤1.5 and a partial prothrombin time (PTT) ≤1.5 times upper limit of normal
  2. For patients on full dose warfarin, in range International Normalized Ratio (usually between 2 and 3) and
  3. Partial prothrombin time (PTT) <1.2 times upper limit of normal
  4. Candidate for administration of postoperative standard platinum-based combination systemic chemotherapy (adequate bone marrow, renal, hepatic function, and blood coagulation parameters)

Exclusion Criteria:

* Any prior treatment modality for the diagnosis of ovarian, fallopian tube, or primary peritoneal cancerPrior surgical attempt of cytoreductive surgery
* Stage I/II disease
* Presence of other invasive malignancies or evidence of other cancer within the past 3 years
* Known active acute hepatitis and confirmed diagnosis of HIV
* Active systemic infection that requires use of parenteral antibiotics
* History of acute coronary syndromes (ACS), within the last 6 months, according to AHA definitions
* New York Heart Association (NYHA) Class II or higher congestive heart failure according to American Heart Association (AHA) definitions
* Canadian Cardiovascular Society (CCS) Class II or higher angina grade according to AHA definitions
* Uncontrolled hypertension defined as > 140/90 and not cleared for surgery at time of consent by cardiologist
* History of cerebral artery disease and prior stroke according to AHA definitions in the last 6 months
* Renal insufficiency with serum creatinine level ≥1.5 times the upper limit of normal or calculated creatinine clearance <60 ml/min
* Patients with concurrent severe medical problems unrelated to malignancy that will preclude compliance with the study or places at an unacceptable risk for participation in the study determinate by study investigators
* Pregnant women are excluded from this study because carboplatin is category D agent with the potential of teratogenic effects. Due to potential risk for adverse events in nursing infants secondary to treatment of the mother with carboplatin, breastfeeding should be discontinued
* Life expectancy of < 12 weeks

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2027-08 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Post-operative complication rates | 30 days post-operative
  Compare post-operative complication rates between study arms

SECONDARY OUTCOMES:
Assessment of quality of life | Baseline, 4 weeks post-operative, upon completion of systemic chemotherapy, and years 1, 2, 3, 4, & 5
  FACT-O questionnaire to assess quality of life in both study arms
Evaluate the rate of progression free survival | at 24 months
  Time from intervention to disease recurrence
Evaluate overall survival | at 1, 3, and 5 years
  Time from intervention to death

OTHER OUTCOMES:
Risk factors for morbidity and mortality | During & at study completion
  Determine percent of patients wtih Grade I-V adverse events according to NCI criteria, Common Terminology Criteria for AE (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Diaz-Montes, M.D., Principal Investigator — Mercy Medical Center; Armando Sardi, M.D., Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States